CLINICAL TRIAL: NCT02111889
Title: Measurement of Tumor Kinase Inhibitor Concentrations Using PET Imaging in Patients With Advanced Solid Malignancies
Brief Title: Tumor Kinase Inhibitor Concentrations Measured by PET
Acronym: PIKTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. MD PhD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012/478; 2012-004961-42 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-11 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Disseminated Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one (Experimental)
  Interventions: Other: [11C] kinase inhibitor PET [15O]water PET and tumor biopsies.

INTERVENTIONS:
Other: [11C] kinase inhibitor PET [15O]water PET and tumor biopsies. — [11C] kinase inhibitor PET (i.e. sorafenib and erlotinib in this study, with the aim to investigate others in future studies) and [15O]water PET will be performed before and after 2 weeks of treatment. Tumor biopsies will be performed before and after 2 weeks of therapy.

SUMMARY:
The investigators hypothesize that response to kinase inhibitors is dependent on achieving pharmacological active drug levels in tumor tissue and that quantitative PET imaging can predict kinase inhibitors tumor concentrations. The ultimate aim is to develop a quantitative PET based imaging tool to differentiate between patients who will respond to therapy with kinase inhibitors.

The main objective of this study is to determine whether tumor concentrations of kinase inhibitors at pharmacological active doses can be predicted from PET studies using tracer amounts (microdosing) of corresponding radiolabeled kinase inhibitors. This objective includes the development and validation of pharmacokinetic models for radiolabeled kinase inhibitors as well as validation of the microdosing concept for kinase inhibitors.

DETAILED DESCRIPTION:
Rationale: Multiple agents targeting specific signaling proteins important for tumor growth and angiogenesis, including (tyrosine) kinase inhibitors and monoclonal antibodies, have been developed and have reached clinical approval. In general, however, these targeted agents induce a response only in a subgroup of cancer patients, while all are exposed to potential toxic therapies. Prior to treatment, it is unknown which patients will respond and why kinase inhibitors are only effective in some, but not all, patients. Clearly, there is a need for a non-invasive in vivo technique to identify those patients who may benefit from treatment with a specific drug.

Positron emission tomography (PET) is a non-invasive technique that enables quantitative measurements of molecular pathways and interactions with picomolar sensitivity and, as such, it has the potential to fulfill the need mentioned above. We expect that response to kinase inhibitors is dependent on achieving active drug levels in tumor tissue. Currently, intratumoral kinase inhibitor levels are being investigated at our institution (ICK study). However, these measurements require fresh tumor biopsies. We hypothesize that radiolabeled kinase inhibitor PET imaging can quantify concentrations of labeled drug in tumor lesions, thereby avoiding burdensome biopsies in the future.

Objective: The main objective of this study is to determine whether tumor concentrations of kinase inhibitors at pharmacological active doses can be predicted from PET studies using tracer amounts (microdosing) of corresponding radiolabeled kinase inhibitors. This objective includes the development and validation of pharmacokinetic models for radiolabeled kinase inhibitors as well as validation of the microdosing concept for kinase inhibitors.

The secondary objectives include exploration whether kinase inhibitor kinetics depend on perfusion (as measured by [15O]water PET) or size (as measured by diagnostic CT/MRI) of tumor lesions, to investigate the presence of a sink that accumulates kinase inhibitor, and to investigate (in)activation of key pathways targeted by the specific kinase inhibitor.

Study design: Single center, non-randomized, interventional proof of concept study.

Study population: Adult patients with advanced, biopsy accessible tumors for whom standard palliative treatment with the kinase inhibitor investigated in this study, i.e. erlotinib and sorafenib, is indicated.

Intervention: Patients will be treated with the kinase inhibitor according to standard treatment. [11C] kinase inhibitor PET (i.e. sorafenib and erlotinib in this study, with the aim to investigate others in future studies) and [15O]water PET will be performed before and after two weeks of treatment. Tumor biopsies will be performed before and during therapy.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Enrollment in this study will require two tumor biopsies, 2x [11C] kinase inhibitor PET, 2x [15O]water PET and arterial blood sampling. The biopsies may cause physical discomfort. During therapy, follow-up will include standard laboratory analysis as well as regular visits to the outpatient clinic. The radiation exposure is acceptable. Patients treated with a kinase inhibitor as standard therapy may benefit from disease regression or stabilization as it has proven clinical benefit in the patient population under investigation. The results of this kinase inhibitor PET imaging study will be strongly supportive for the development of non-invasive, personalized treatment strategies thereby avoiding 1) cumbersome tumor biopsies, 2) unwanted exposure to potentially toxic drugs and 3) costly therapy without clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically confirmed diagnosis of an advanced or metastatic solid malignancy.
2. Patients must have confirmed radiological or clinical progressive disease.
3. Patients must have at least one measurable tumor lesion outside the liver.
4. Indication for standard use of sorafenib or erlotinib
5. Age ≥ 18 years.
6. ECOG Performance Status ≤ 2.
7. Life expectancy of at least 12 weeks.
8. Patients should be able to swallow oral medication.
9. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   1. Hemoglobin > 6.0 mmol/L
   2. Absolute neutrophil count (ANC) >1,5 x 10*9/L
   3. Platelet count ≥ 100 x 10*9/L
   4. Total bilirubin < 2 times the upper limit of normal (ULN)
   5. ALT and AST < 2.5 x ULN; < 5x ULN in case of liver metastases, except for patients with hepatocellular carcinoma, than Child Pugh classification A-B.
   6. Alkaline phosphatase < 4 x ULN; < 5x ULN in case of liver metastases, except for patients with hepatocellular carcinoma, than Child Pugh classification A-B.
   7. Serum creatinine eGFR ≥ 50 mL/min.
   8. PT-INR/PTT < 1.5 x ULN, unless coumarin derivatives are used.
   9. Activated partial thromboplastin time < 1.25 x ULN (therapeutic anticoagulation therapy is allowed, if this treatment can be interrupted for a biopsy as judged by the treating physician).

Exclusion Criteria:

1. Concurrent treatment with other anticancer agents or experimental drugs.
2. History of cardiac disease:

   1. Congestive heart failure >NYHA class 2.
   2. Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening).
   3. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
3. Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 2 separate measurements.
4. Uncontrolled infections (> grade 2 NCI-CTC version 4.0).
5. Subjects with serious non-healing wound, ulcer, or bone fracture.
6. Patients with thromboembolic events within 3 months prior to study inclusion.
7. Significant skin condition interfering with treatment
8. Patients undergoing renal dialysis.
9. Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must agree to use adequate barrier birth control measures (e.g., cervical cap, condom, or diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between study drug and oral contraceptives. Concomitant use of oral and barrier contraceptives is advised. Contraception is necessary for at least 6 months after receiving the study kinase inhibitor.
10. Concomitant use of dexamethasone, anti-convulsants and anti-arrhythmic drugs other than digoxin or beta blockers.
11. Major surgery within 28 days prior to start of treatment.
12. Medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
13. Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
tumor concentrations of a microdose radiolabeled kinase inhibitor | before start of treatment and after two weeks of treatment with a kinase inhibitor
  a radiolabeled kinase inhibitor PET is used to asses this outcome measure
tumor concentrations of therapeutic kinase inhibitor | after 2 weeks of treatment with a kinase inhibitor
  measured in a tumor biopsy with LC-MS/MS

SECONDARY OUTCOMES:
tumor perfusion | before treatment and after two weeks of treatment with a kinase inhibitor
  measured with [15O]H2O PET
tumor size | before treatment and after two months of treatment
  Measured with CT
(in)activation of key pathways targeted by the specific kinase inhibitor | after two weeks of treatment with a kinase inhibitor
  immunohistochemical stainings, Western blotting, phosphoproteomics

CONTACTS AND LOCATIONS:
Overall Officials: H. M. Verheul, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Bahce I, Smit EF, Lubberink M, van der Veldt AA, Yaqub M, Windhorst AD, Schuit RC, Thunnissen E, Heideman DA, Postmus PE, Lammertsma AA, Hendrikse NH. Development of [(11)C]erlotinib positron emission tomography for in vivo evaluation of EGF receptor mutational status. Clin Cancer Res. 2013 Jan 1;19(1):183-93. doi: 10.1158/1078-0432.CCR-12-0289. Epub 2012 Nov 7. PMID 23136193